CLINICAL TRIAL: NCT00706030
Title: A Phase 1/2 Study Of HKI-272 In Combination With Vinorelbine In Subjects With Solid Tumors And Metastatic Breast Cancer
Brief Title: Study Evaluating Neratinib (HKI-272) In Combination With Vinorelbine In Subjects With Solid Tumors And Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3144A1-2204 / B1891015
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer; Advanced Malignant Solid Tumors
Keywords: Metastatic breast cancer; HKI-272; Neratinib; Nerlynx; PB-272
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- neratinib 160 mg + vinorelbine (Experimental): neratinib 160 mg tablets administered daily by mouth, vinorelbine 25 mg/m^2 administered IV on day 1 and day 8 of 21 day cycle
  Interventions: Drug: neratinib; Drug: vinorelbine
- neratinib 240 mg + vinorelbine (Experimental): neratinib 240 mg tablets administered daily by mouth, vinorelbine 25 mg/m^2 administered IV on day 1 and day 8 of 21 day cycle
  Interventions: Drug: neratinib; Drug: vinorelbine
- neratinib 240 mg + vinorelbine, No Prior Lapatinib (Experimental): neratinib 240 mg tablets administered daily by mouth, vinorelbine 25 mg/m^2 administered IV on day 1 and day 8 of 21 day cycle
  Interventions: Drug: neratinib; Drug: vinorelbine
- neratinib 240 mg + vinorelbine, Prior Lapatinib (Experimental): neratinib 240 mg tablets administered daily by mouth, vinorelbine 25 mg/m^2 administered IV on day 1 and day 8 of 21 day cycle
  Interventions: Drug: neratinib; Drug: vinorelbine

INTERVENTIONS:
Drug: neratinib
  Other Names: HKI-272; Nerlynx
Drug: vinorelbine

SUMMARY:
The purpose of this study is to identify the highest tolerable dose of neratinib (HKI-272) in combination with vinorelbine and to assess the safety of the combination of the two drugs as well as to obtain preliminary information on whether the combination of the two drugs has any effect on solid tumors.

The study will be conducted in two parts. In the first part, testing will be done on up to 12 subjects to determine the highest tolerable dose of HKI-272 and vinorelbine in patients with advanced solid tumors. In the second part of the study, approximately 60 additional subjects with metastatic ErbB-2-positive breast cancer, with no prior exposure to lapatinib, are planned to be added to better define the tolerability and preliminary activity of HKI-272 in combination with vinorelbine. Up to 20 additional subjects with ErbB-2-positive breast cancer with prior lapatinib exposure are also planned to be enrolled in part 2 for exploratory analyses.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pathologic diagnosis of a solid tumor that is not curable with available therapies for which HKI-272 plus vinorelbine is a reasonable treatment option (part 1 only) or Confirmed pathologic diagnosis of ErbB-2-positive breast cancer (current stage IV) in female subjects for which vinorelbine plus HKI-272 is a reasonable treatment option (part 2 only).
* At least 1 prior antineoplastic chemotherapy treatment regimen for metastatic disease and at least 1 prior treatment with a trastuzumab-containing regimen for at least 6 weeks, for metastatic disease or subject relapsing under adjuvant treatment (part 2 only).
* At least 1 measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST).

Exclusion Criteria:

* More than 2 prior antineoplastic treatment regimens (excluding hormonotherapy) for metastatic disease. Subjects who relapsed under adjuvant treatment shouldn't have received more than one line of chemotherapy for metastatic disease (part 2 only).
* Prior treatment with vinorelbine for metastatic setting, or prior treatment with any ErbB-2 targeted agents except trastuzumab (part 2 only). Up to 20 subjects with ErbB-2-overexpressing metastatic breast cancer who have been previously exposed to lapatinib but are not refractory to lapatinib may be enrolled in part 2.
* Prior treatment with anthracyclines with a cumulative dose of doxorubicin of greater than 400 mg/m2, or of epirubicin dose of greater than 800 mg/m2, or the equivalent dose for other anthracyclines or derivatives (part 2 only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-04-29 (Actual); Primary Completion 2009-10 (Actual); Study Completion 2018-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (35):
- United States (8):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - Norris Cotton Cancer Center, Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Medical Center, New York, New York
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - Albert Einstein Cancer Center, The Bronx, New York
  - Carolinas Hematology-Oncology Associates, Charlotte, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Belgium (3):
  - AZ Klina Brasschaat, Brasschaat
  - Institut Jules Bordet, Brussels
  - St.-Augustinus Hospital Oncology Department, Wilrijk
- China (4):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The Hospital Affiliated Academy Military Medical Science, Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
- France (4):
  - Centre Paul Papin, Angers
  - Institut Paoli Calmette, Marseille
  - Institut Curie, Département d'Oncologie Médicale, Paris
  - Institut Claudius Regaud, Toulouse
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - UNIMED Medical Institute, Hong Kong
- Martini Ziekenhuis / Afdeling Interne Geneeskunde, Groningen, Netherlands
- Poland (2):
  - Centrum Onkologii Ziemii Lubelskiej, Oddział Chemioterapii, Lublin
  - Wojskowy Instytut Medyczny, Klinika Onkologii, Warsaw
- Spain (4):
  - Centro Oncologico de Galicia, A Coruña
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Arnau de Vilanova, Servicio de Oncologia Medica, Lleida
  - Hospital 12 de Octubre, Servicio de Oncologia Medica, Madrid
- Onkologiska Kliniken Universitetssjukhuset i Lund, Lund, Sweden
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (5):
  - Broomfield Hospital, Chelmsford, Essex
  - Southampton General Hospital, Southampton, Hampshire
  - Christie NHS Foundation Trust, Manchester, Lancashire
  - Velindre Cancer Centre, Cardiff
  - Guy's and St. Thomas' NHS Foundation Trust, Guy's Hospital, London

REFERENCES:
- [Derived] Awada A, Dirix L, Manso Sanchez L, Xu B, Luu T, Dieras V, Hershman DL, Agrapart V, Ananthakrishnan R, Staroslawska E. Safety and efficacy of neratinib (HKI-272) plus vinorelbine in the treatment of patients with ErbB2-positive metastatic breast cancer pretreated with anti-HER2 therapy. Ann Oncol. 2013 Jan;24(1):109-16. doi: 10.1093/annonc/mds284. Epub 2012 Sep 11. PMID 22967996

RESULTS

PARTICIPANT FLOW:
Groups:
- Neratinib 160 mg + Vinorelbine 25 mg/m²: Neratinib 160 mg qd + Vinorelbine 25 mg/m² IV on days 1 and 8 every 3 weeks
- Neratinib 240 mg + Vinorelbine 25 mg/m²: Neratinib 240 mg qd + Vinorelbine 25 mg/m² IV on days 1 and 8 every 3 weeks
- Neratinb 240 mg + Vinorelbine 25 mg/m² - No Prior Lapatinib: Neratinib 240 mg qd + Vinorelbine 25 mg/m² IV on days 1 and 8 every 3 weeks, with no prior lapatinib exposure
- Neratinib 240 mg + Vinorelbine 25 mg/m² - Prior Lapatinib: Neratinib 240 mg qd + Vinorelbine 25 mg/m² IV on days 1 and 8 every 3 weeks, with prior Lapatinib exposure
Period: Overall Study
Arm/Group | Neratinib 160 mg + Vinorelbine 25 mg/m² | Neratinib 240 mg + Vinorelbine 25 mg/m² | Neratinb 240 mg + Vinorelbine 25 mg/m² - No Prior Lapatinib | Neratinib 240 mg + Vinorelbine 25 mg/m² - Prior Lapatinib
Started | 6 | 6 | 64 | 16
Treated | 6 | 6 | 64 | 15
Completed | 0 | 0 | 4 | 0
Not Completed | 6 | 6 | 60 | 16
Not completed — Disease Progression | 4 | 6 | 46 | 12
Not completed — Adverse Event | 1 | 0 | 4 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 0
Not completed — Not recorded | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Failed to return | 0 | 0 | 1 | 0
Not completed — Symptomatic Deterioration | 0 | 0 | 1 | 0
Not completed — No treatment received | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neratinib 160 mg + Vinorelbine 25 mg/m² | Neratinib 240 mg + Vinorelbine 25 mg/m² | Neratinb 240 mg + Vinorelbine 25 mg/m² - No Prior Lapatinib | Neratinib 240 mg + Vinorelbine 25 mg/m² - Prior Lapatinib | Total
Number analyzed (Participants) | 6 | 6 | 64 | 15 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (14.8) | 54.3 (13.9) | 51.1 (10.6) | 52.1 (9.8) | 51.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 64 | 15 | 89
  Male | 0 | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 18 | 6 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 2
  White | 4 | 5 | 43 | 9 | 61
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall Response Rate (ORR), subjects with CR or PR by independent review in subjects with ErbB-2-positive breast cancer treated at the MTD of neratinib in combination with vinorelbine per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.0: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Non-PD for non-target lesions, and no new lesions.
Time Frame: From first dose date to progression or last tumor assessment, up to four years and six months.
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinb 240 mg + Vinorelbine 25 mg/m² - No Prior Lapatinib | Neratinib 240 mg + Vinorelbine 25 mg/m² - Prior Lapatinib
Number analyzed (Participants) | 64 | 15
percentage of participants | 35.9 [24.3 to 48.9] | 13.3 [1.7 to 40.5]

2. Secondary Outcome: Clinical Benefit Rate
Description: Percentage of participants with partial response (PR) or complete response (CR) or stable disease > 24 weeks by independent assessment for subjects with ErbB-2-positive breast cancer treated at the MTD of neratinib in combination with vinorelbine, per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v.1.0: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Non-PD for non-target lesions, and no new lesions.
Time Frame: From first dose date to progression or last tumor assessment, up to four years and six months.
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinb 240 mg + Vinorelbine 25 mg/m² - No Prior Lapatinib | Neratinib 240 mg + Vinorelbine 25 mg/m² - Prior Lapatinib
Number analyzed (Participants) | 64 | 15
percentage of participants | 64.1 [51.1 to 75.7] | 40.0 [16.3 to 67.7]

3. Secondary Outcome: Progression-Free Survival
Description: Number of weeks between the date of the first dose of test article and the first date of disease recurrence or progression, or death due to any cause, was documented, censored at the last evaluation, investigator assessment. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (v1.0), as at least a 20% increase in the sum of the longest diameters (LD) of target lesions, taking as reference the nadir LD, meaning the smallest sum of the LDs recorded since the treatment started; or unequivocal progression of existing nontarget lesions; or the appearance of any new lesions.
Time Frame: From first dose date to progression or death, up to four years and six months.
Population: Evaluable population, independent assessment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Neratinb 240 mg + Vinorelbine 25 mg/m² - No Prior Lapatinib | Neratinib 240 mg + Vinorelbine 25 mg/m² - Prior Lapatinib
Number analyzed (Participants) | 56 | 12
weeks | 48.0 [30.9 to 65.1] | 22.7 [12.0 to 41.0]

4. Secondary Outcome: Duration Of Response
Description: Duration of response for subjects who had complete or partial response from first response to disease progression, death or last assessment per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.0: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Non-PD for non-target lesions, and no new lesions.
Time Frame: From start date of response to first PD/death, up to four years and six months.
Population: Subjects in evaluable population who had CR or PR according to Independent Assessment.
Measure: Median (Full Range); unit: weeks
Groups:
- Neratinib 20 mg + Vinorelbine 25 mg/m² - Prior Lapatinib: Neratinib 240 mg qd + Vinorelbine 25 mg/m² IV on days 1 and 8 every 3 weeks, with prior Lapatinib exposure.
Arm/Group | Neratinb 240 mg + Vinorelbine 25 mg/m² - No Prior Lapatinib | Neratinib 20 mg + Vinorelbine 25 mg/m² - Prior Lapatinib
Number analyzed (Participants) | 23 | 1
weeks | 52.7 [11.6 to 96.1] | 77.7 [77.7 to 77.7]

5. Primary Outcome: Maximum Tolerated Dose
Description: Maximum Tolerated Dose (MTD) of Neratinib in combination with vinorelbine in subjects with advanced solid tumors.
Time Frame: From Day 1 to Day 21.
Population: Safety population of Study Part 1. Treated set including patients eligible for MTD determination.
Measure: Number; unit: mg
Groups:
- Part 1: Maximum Tolerated Dose (MTD) of neratinib, daily, in combination with Vinorelbine 25 mg/m2 IV on days 1 and 8 every 3 weeks, associated with the dose limiting toxicity data.
Arm/Group | Part 1
Number analyzed (Participants) | 12
mg | 240

ADVERSE EVENTS:
Time Frame: From first dose through 28 days after last dose, up to four years and six months.
Arm/Group | Neratinib 160 mg + Vinorelbine 25 mg/m² | Neratinib 240 mg + Vinorelbine 25 mg/m² | Neratinb 240 mg + Vinorelbine 25 mg/m² - No Prior Lapatinib | Neratinib 240 mg + Vinorelbine 25 mg/m² - Prior Lapatinib
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 21/64 | 5/15
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 64/64 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib 160 mg + Vinorelbine 25 mg/m² (N=6) | Neratinib 240 mg + Vinorelbine 25 mg/m² (N=6) | Neratinb 240 mg + Vinorelbine 25 mg/m² - No Prior Lapatinib (N=64) | Neratinib 240 mg + Vinorelbine 25 mg/m² - Prior Lapatinib (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 4 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ureteric haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Mastectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib 160 mg + Vinorelbine 25 mg/m² (N=6) | Neratinib 240 mg + Vinorelbine 25 mg/m² (N=6) | Neratinb 240 mg + Vinorelbine 25 mg/m² - No Prior Lapatinib (N=64) | Neratinib 240 mg + Vinorelbine 25 mg/m² - Prior Lapatinib (N=15)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 15 | 5
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 21 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 36 | 9
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 5 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 5 | 0
Eye irritation (Eye disorders) | 0 | 1 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Scleral haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 5 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 22 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 8 | 3
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 5 | 10 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 6 | 61 | 15
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 5 | 0
Gingival ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 6 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 10 | 2
Nausea (Gastrointestinal disorders) | 4 | 3 | 35 | 7
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 8 | 2
Tongue discolouration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 24 | 10
Asthenia (General disorders) | 0 | 2 | 16 | 5
Chest discomfort (General disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 3 | 3 | 24 | 4
Influenza like illness (General disorders) | 0 | 0 | 5 | 1
Malaise (General disorders) | 0 | 0 | 4 | 2
Medical device complication (General disorders) | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 12 | 1
Oedema peripheral (General disorders) | 0 | 1 | 7 | 1
Pain (General disorders) | 1 | 0 | 2 | 1
Pyrexia (General disorders) | 0 | 1 | 19 | 2
Thrombosis in device (General disorders) | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 3 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1 | 9 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 3 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 7 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1
Spinal cord infection (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 7 | 1
Urinary tract infection (Infections and infestations) | 1 | 2 | 6 | 3
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase (Investigations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 12 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 9 | 4
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2 | 2
Haemoglobin decreased (Investigations) | 0 | 0 | 4 | 1
High density lipoprotein decreased (Investigations) | 0 | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1
Red blood cells urine (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 4 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 5 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 20 | 7
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 4 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 5 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 6 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 7 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 12 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 10 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 11 | 3
Dysgeusia (Nervous system disorders) | 2 | 1 | 6 | 0
Headache (Nervous system disorders) | 2 | 2 | 18 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 5 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 9 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 5 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 9 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 2 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 5 | 0
Depression (Psychiatric disorders) | 0 | 1 | 3 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 5 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 4 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 2 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ureteric haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 2 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 13 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 7 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 5 | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 12 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 7 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 10 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 2 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less